CLINICAL TRIAL: NCT03874078
Title: Turkish Version of Kids-BESTest (Balance Evaluation Systems Test) and Kids-Mini-BESTest, Validity and Reliability for School-Aged Children
Brief Title: Turkish Version of Kids BESTest, Validity and Reliability for School-Aged Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Sema BÜĞÜŞAN ORUÇ, Principal Investigator, Ordu University
Other Study IDs: ORDU346
Record Dates: First submitted 2019-03-11; First posted 2019-03-14 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Children, Only; Adolescent
Keywords: school children; balance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to present the Turkish version of Kids-BESTest and Kids-Mini-BESTest and practice of validity and reliability on school-aged children will be performed by utilizing the Turkish version of Kids-BESTest and Kids-Mini-BESTest in this study.

DETAILED DESCRIPTION:
Postural control is the ability to control the body position in space for the purpose of postural stability.

Full-Balance Evaluation Systems Test (BESTest) comprises 36 items and evaluate all components of postural control. Full-BESTest classifies postural control across six domains as: Biomechanical constraints, Stability Limits/Verticality, Transitions - Anticipatory Postural Adjustment, Reactive Postural Response, Sensory Orientation and Stability in Gait. Items in each domain are scored from 0 (worst performance) to 3 (best performance), all requires 30 minutes (maximum score is 108).

Because of the clinical time limits, MiniBESTest is a shortened version of BESTest was developed with 14 tasks. MiniBESTest still addresses almost all components of postural control and can be performed 15 min. MiniBESTest is one of the most common methods practiced for adult patients. Recently BESTest and miniBESTest had modified by Dewar et al for 8-14 aged children which termed Kids-BESTest and Kids-Mini-BESTest.

The aim of this study is to present the Turkish version of Kids-BESTest and Kids-Mini-BESTest and practice of validity and reliability on school-aged children will be performed by utilizing the Turkish version of Kids-BESTest and Kids-Mini-BESTest in this study.

ELIGIBILITY:
Inclusion Criteria:

* Typical developing school-aged children who are volunteers.

Exclusion Criteria:

* Has medical or behavioural disorders

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Typical developing school-aged children (8-14 years)
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-05-06 (Estimated); Primary Completion 2021-11-04 (Estimated); Study Completion 2022-01-02 (Estimated)

PRIMARY OUTCOMES:
Kids BESTest | 30 minutes.
  Kids-BESTest has 36 items and six domains as: Biomechanical constraints, Stability Limits/Verticality, Transitions - Anticipatory Postural Adjustment, Reactive Postural Response, Sensory Orientation and Stability in Gait.
  Items in each domain are scored from 0 (worst performance) to 3 (best performance) with maximum score of 108.
Kids Mini- BESTest | 15 minutes
  It has 14 items and four domains as Anticipatory Postural Adjustments, Reactive Postural Response, Sensory Orientation and Stability in Gait, to focus on the construct of 'dynamic balance'. Mini-BESTest is scored from 0 (worst performance) to 2 (best performance) with a maximum of 28 points.
The Four Square Step Test (FSST) | 3minutes
  The Four Square Step Test (FSST) is a clinical test that assesses balance in the presence of task and environmental constraints. The FSST measures the time an individual takes to step rapidly in four different directions.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dewar R, Claus AP, Tucker K, Ware R, Johnston LM. Reproducibility of the Balance Evaluation Systems Test (BESTest) and the Mini-BESTest in school-aged children. Gait Posture. 2017 Jun;55:68-74. doi: 10.1016/j.gaitpost.2017.04.010. Epub 2017 Apr 6. PMID 28419876
- [Background] Dewar R, Claus AP, Tucker K, Ware RS, Johnston LM. Reproducibility of the Kids-BESTest and the Kids-Mini-BESTest for Children With Cerebral Palsy. Arch Phys Med Rehabil. 2019 Apr;100(4):695-702. doi: 10.1016/j.apmr.2018.12.021. Epub 2019 Jan 9. PMID 30639271
- [Background] Horak FB, Wrisley DM, Frank J. The Balance Evaluation Systems Test (BESTest) to differentiate balance deficits. Phys Ther. 2009 May;89(5):484-98. doi: 10.2522/ptj.20080071. Epub 2009 Mar 27. PMID 19329772